CLINICAL TRIAL: NCT04192968
Title: Follow-up of Cochlear Implanted Children at 3 Years : Comparison of Electrophysiological and Speech-language Results
Acronym: ImplantHear3
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190839; 2019-A02402-55 (Other: ID RCB number)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cochlear Implantation
Keywords: Cochlear implantation; Automated cortical auditory evoked potentials; Speech-language therapy; Children; Cortical auditory evoked potentials; Electrical potentials via the implant
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Children implanted cochlear since 3 years in uni or bilateral and followed in the pediatric otolaryngology department of Necker-Enfants Malades Hospital.
  Interventions: Other: Cortical auditory evoked potentials
- Patients with disappointing language development or poor cortical responses: Children having participated in the main ImplantHear3 study and who present with disappointing language development or poor cortical responses.
  Interventions: Other: Additional exams

INTERVENTIONS:
Other: Cortical auditory evoked potentials — Recording of automated cortical auditory evoked potentials in response to a vocal stimulus.
  Groups: Patients
Other: Additional exams — * Cortical auditory evoked potentials Recording of automated cortical auditory evoked potentials in response to a vocal stimulus.
  * Recording of cortical auditory evoked potentials in response to a click
  * Realization of electrical potentials via the implant Followed up once a year during a visit scheduled for usual care, for 3 years, that to say up to 6 years post-implant.
  Groups: Patients with disappointing language development or poor cortical responses

SUMMARY:
The objective of the study is to compare the responses recorded with automated cortical auditory evoked potentials, of children who had one or two cochlear implants for 3 years, and the results of the speech therapy assessment.

24 patients in the main ImplantHear3 study presented with disappointing language development or poor cortical responses. These patients will be followed up once a year, during a visit scheduled for the usual care, until 6 years post-implant, in order to make it possible to objectify the quality of the auditory rehabilitation received by the child.

DETAILED DESCRIPTION:
Children with severe to profound deafness can benefit from cochlear rehabilitation, combined with a speech-language therapy. At present, 70 to 80% of children with congenital - profound deafness who are implanted at an early age will have a language level identical to their hearing peers. But 20 to 30% of them will be able to present linguistic difficulties.

The objective recording of the cortical activity in response to a sound stimulus gives a proof of the quality of the auditory stimulation that is perceived by the cortex, an essential condition for the further linguistic development of the child. By the use of complex stimuli of speeching type, all the channels involved in the auditory processing are analyzed.

The recording in routine clinical practice of the cortical auditory evoked potentials in response to a vocal stimulus makes it possible to objectify the quality of the auditory rehabilitation received by the child.

The implanted children all benefit from regular and prolonged speech therapy follow-up, with a complete evaluation every year. It is important to regularly monitor the linguistic evolution of young children who are implanted in order to identify children at risk of poorer linguistic development at an early age.

The objective of the study is to compare the responses recorded with automated cortical auditory evoked potentials, of children who had one or two cochlear implants for 3 years, and the results of the speech therapy assessment.

24 patients in the main ImplantHear3 study presented with disappointing language development or poor cortical responses. These patients will be followed up to 6 years post-implant by carrying out, during a visit scheduled for patient care, once a year for 3 years:

* Recording of automated cortical auditory evoked potentials in response to a vocal stimulus, as performed for the main study, but also :
* Recording of cortical auditory evoked potentials in response to a click
* Realization of electrical potentials via the implant And this in order to make it possible to objectify the quality of the auditory rehabilitation received by the child.

The objectives of the ancillary study are :

Comparison of the responses recorded to automated cortical auditory evoked potentials, of children who have had one or two cochlear implants for 4 years, with the results of speech therapy and up to 6 years post-implant.

Look for prognostic factors of poor linguistic development: correlate the electrophysiological results, the adjustment parameters, the modalities of hearing rehabilitation, the side of the cochlear implantation, and the audiometric thresholds with the results of the speech therapy assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 42 months to 17 years on the day of inclusion.
* Patient who has received one or two cochlear implants between August 1, 2016 and November 1, 2017 and after 3 years of follow-up for the first implant.
* Non-opposition of the holders of the parental authority and the patient.

Exclusion Criteria:

* Patients over 15 years of age at implantation.
* Patient relocated between August 1, 2016 and November 1, 2017.

Ages: 42 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children implanted for 3 years, in unilateral or bilateral and followed in the pediatric otolaryngology department of the Necker-Enfants Malades Hospital in Paris.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
Automated cortical auditory evoked potentials results | Annual assessment performed during 3 years.
  Latency and amplitude of the waves P1, N1, P2, N2.
Speech therapy result | Annual assessment performed during 3 years.
  Percentage of recognition Open Set Words :
  * cochlear implant 1,
  * cochlear implant 2,
  * 2 cochlear implants together,
  * cochlear implant and hearing aid together.

SECONDARY OUTCOMES:
Value of p (HearLab) | Annual assessment performed during 3 years.
  Analysis of the automatic validation by HearLab: value of p, for each vocal stimulus / m /, / g /, / t /, and / s / as a function of the intensity : 55, 65, 75 Db.
Latencies P1, N1, P2, N2 (HearLab) | Annual assessment performed during 3 years.
  Study of the latencies P1, N1, P2, N2 by HearLab, as a function of the stimulus / m /, / g /, / t /, and / s /, intensity : 55, 65, 75 dB and age.
Amplitudes P1, N1, P2, N2 (HearLab) | Annual assessment performed during 3 years.
  Study of the amplitudes P1, N1, P2, N2 by HearLab, as a function of the stimulus / m /, / g /, / t /, and / s /, intensity : 55, 65, 75 dB and age.
Setting parameters | Annual assessment performed during 3 years.
  Active electrode number, minimum thresholds and comfort, dynamic, on each side, pulse width and frequency.
Auditory rehabilitation | Annual assessment performed during 3 years.
  - Type of auditory rehabilitation : uni or bilateral cochlear implant : if bilateral cochlear implant : sequential or simultaneous, if unilateral cochlear implant : side, contralateral hearing aid (yes or no),
  * age at implantation (for each side if bilateral)
  * cochlear implant Device
  * electrode
  * datalogging for each cochlear implant : never/ <6 hours/ 6-9hours/>10 hours,
  * hearing aid device.
Residual hearing level | Annual assessment performed during the year of the 3 years following cochlear implantation.
  Auditory level without devices :
  right Ear : 250, 500, 1000, 2000, 4000 Hz, left Ear : 250, 500, 1000, 2000, 4000 Hz.
Deafness characteristics | Annual assessment performed during the year of the 3 years following cochlear implantation.
  * age at the diagnosis,
  * age at the beginning of deafness,
  * etiology of the deafness,
  * syndromic deafness or not.
Latencies P1, N1, P2, N2 | Annual assessment performed during 3 years.
  Study of the latencies P1, N1, P2, N2 by cortical auditory evoked potentials results (in response to click)
Amplitudes P1, N1, P2, N2 | Annual assessment performed during 3 years.
  Study of the amplitudes P1, N1, P2, N2 by cortical auditory evoked potentials results (in response to click)
Latency study of the wave V | Annual assessment performed during 3 years.
  Electrical evoked potentials results via the implant
Amplitude study of the wave V | Annual assessment performed during 3 years.
  Electrical evoked potentials results via the implant
Stimulation level and pulse duration required to generate a wave V | Annual assessment performed during 3 years.
  Electrical evoked potentials results via the implant

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Loundon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Isabelle Rouillon, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No